CLINICAL TRIAL: NCT00897221
Title: An Open-label, Single Treatment, Safety and Efficacy, Long-term Study of Deferiprone in Subjects With Friedreich's Ataxia
Brief Title: A Study Investigating the Long-term Safety and Efficacy of Deferiprone in Patients With Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Dian Shaw, ApoPharma Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LA29-EXT
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose 1 (Experimental): Deferiprone oral solution 20 mg/kg/day
  Interventions: Drug: Deferiprone oral solution 100mg/mL
- Dose 2 (Experimental): Deferiprone oral solution 40 mg/kg/day
  Interventions: Drug: Deferiprone oral solution 100 mg/mL

INTERVENTIONS:
Drug: Deferiprone oral solution 100mg/mL — Deferiprone oral solution (20 mg/kg/day)
  Other Names: Ferriprox
  Arms: Dose 1
Drug: Deferiprone oral solution 100 mg/mL — Deferiprone oral solution(40mg/kg/day)
  Other Names: Ferriprox
  Arms: Dose 2

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of deferiprone in subjects with Friedreich's ataxia (FRDA).

The secondary objective is to evaluate the long-term efficacy of deferiprone for the treatment of FRDA.

The tertiary objectives are to evaluate the effect of deferiprone on:

1. cardiac function,
2. quality of life, and
3. functional status.

DETAILED DESCRIPTION:
This is a multi-centre, open-label, non-randomized, single treatment, safety and efficacy study. All subjects who completed the LA29-0207 study are eligible for participation. Participants will receive deferiprone oral solution at the same dose (20 or 40 mg/kg/day) that they were assigned for LA29-0207. The duration of treatment will be 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who completed the ApoPharma study LA29-0207
2. Female subjects of childbearing potential must have a negative pregnancy test.
3. Male subjects must confirm that he and/or his female partner will use an effective method of contraception for the length of the trial and for 30 days following completion of the study or early termination.
4. Signed and witnessed written informed consent/assent, obtained prior to the first study intervention, as well as the ability to adhere to study restrictions, appointments and evaluation schedules.

Exclusion Criteria:

1. Serum Ferritin and Hemoglobin (Hb) levels are below the reference range for age and sex-matched controls.
2. Unable to complete T25FW AND with a score > 5 minutes in the 9HPT. Subjects who can complete T25FW or with a score ≤ 5 minutes in the 9HPT will be allowed to enrol).
3. Doubling of score on 9HPT or T25FW compared to their study baseline results in LA29-0207.
4. History or evidence of neutropenia/agranulocytosis defined by a confirmed absolute neutrophil count (ANC) < 1.5 x 109/L or thrombocytopenia defined by a platelet count <150 x 109/L.
5. Occurrence of SAEs or any other AEs during the LA29-0207 study, which in the opinion of the investigator cause the patient's participation in the extension study to be inappropriate.
6. Unable to comply with requirements of the protocol.
7. Pregnant, breastfeeding or planning to become pregnant during the study period.
8. QTc interval >450ms.
9. Have been on antioxidants prior to start of study treatment.

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The patient's long-term tolerance of treatment will be assessed by the occurence of adverse events. | 52 weeks

SECONDARY OUTCOMES:
The long-term efficacy of deferiprone will be assessed. Efficacy measures include the 9HPT, T25FW, LCLA, ICARS and FARS. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Pandolfo, M.D., Principal Investigator — Hospital Erasme, Brussels, Belgium; Arnold Munnich, M.D., Principal Investigator — Hospital Necker-Enfants Malades, Paris, France; Franco Taroni, M.D., Principal Investigator — Fondazione IRCCS Istituto Neurologico "C. Besta", Milan, Italy; Javier Arpa, M.D., Principal Investigator — La Fundaction Para la Investigacion Biomedica, Madrid, Spain
Locations (4):
- Hospital Erasme, Brussels, Belgium
- Hospital Necker-Enfants Malades, Paris, France
- Fondazione IRCCS Istituto Neurologico "C. Besta", Milan, Italy
- La Fundacion Para la Investigacion Biomedica, Madrid, Spain